CLINICAL TRIAL: NCT02678923
Title: A Placebo-controlled, Double-blind, Randomized Trial to Compare the Effect of Treatment on Plaque Burden as Determined by Intravascular Ultrasound and to Evaluate the Efficacy, Pharmacokinetics, Safety, and Tolerability of MDCO-216 Given as Multiple Weekly Infusions in Subjects With a Recent Acute Coronary Syndrome
Brief Title: MDCO-216 Infusions Leading to Changes in Atherosclerosis: A Novel Therapy in Development to Improve Cardiovascular Outcomes - Proof of Concept Intravascular Ultrasound (IVUS), Lipids, and Other Surrogate Biomarkers Trial
Acronym: PILOT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDCO-APO-15-01; 2015-000826-13 (EudraCT Number)
Record Dates: First submitted 2016-02-05; First posted 2016-02-10 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-06

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — MDCO-216; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MDCO-216 (Experimental): 20 mg/kg of MDCO-216 administered intravenously (IV) as a 360 milliliter (mL) infusion over 2 hours on Days 1, 8, 15, 22, and 29
  Interventions: Drug: MDCO-216
- Placebo (Placebo Comparator): 360 mL of placebo (0.9% sodium chloride [NaCl] solution) infusion, IV, over 2 hours on Days 1, 8, 15, 22, and 29
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDCO-216
  Other Names: Recombinant Apo A-I Milano (rApoA-IM)
  Arms: MDCO-216
Drug: Placebo
  Other Names: NaCl Solution
  Arms: Placebo

SUMMARY:
This study will be a proof-of-concept, placebo-controlled, double-blind, randomized trial in participants with a recent acute coronary syndrome (ACS) to evaluate the efficacy, pharmacokinetics, safety, tolerability, disease progression measures by IVUS, and pharmacodynamics of MDCO-216 infusion. Eligible participants will be randomized to receive 5 infusions of MDCO-216 20 milligrams/kilogram (mg/kg) or placebo in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Have experienced a recent ACS event within 14 days of screening that requires a clinically indicated coronary angiogram.
* A qualifying ACS event will be defined as follows: a diagnosis of a qualifying myocardial infarction (MI) event will be defined by abnormal levels of cardiac biomarkers (troponin I or T or creatine kinase myoglobin [CK-MB] mass) with at least one determination greater than the 99th percentile or upper limits of normal (ULN) for the laboratory and at least one of the following: chest discomfort or symptoms of myocardial ischemia (≥10 minutes) at rest within 24 hours prior to hospitalization for MI and/or new electrocardiogram (ECG) findings (or presumed new if no prior ECG available) indicative of acute myocardial ischemia in absence of left ventricular hypertrophy (LVH) and left bundle branch block (LBB).
* Baseline coronary angiogram must meet all of the following criteria for IVUS interrogation of target artery:

  * Target artery must be accessible to the IVUS catheter
  * Target artery must have a stenotic area of ≥20% and <50% in lumen diameter by angiographic visual estimation within the length of the native coronary artery ("target segment") for imaging by IVUS
  * Target artery has not undergone prior percutaneous coronary intervention (PCI) or coronary artery bypass graft surgery (CABG)
  * Target artery is not currently a candidate for intervention or a likely candidate for intervention over the treatment phase of the study and until the second IVUS interrogation at Day 36; the target artery may not be a bypass graft
  * Target artery may not be the culprit vessel for a previous MI.

The target artery may have the following:

* A lesion of up to 60% stenosis, distal to the target segment, provided that this area is not a target for PCI or CABG
* A single branch of the "target vessel" may have a narrowing ≤70% by visual estimation, provided that the branch in question is not a target for PCI or CABG.
* Willing and able to give informed consent before initiation of any study-related procedures and willing to comply with all required study procedures.

Exclusion Criteria:

* Baseline IVUS not completed due to non-qualifying coronary angiogram as demonstrated by a greater than 50% reduction in lumen of the left main coronary artery by visual estimation, or extensive coronary artery disease (CAD) with no target vessel for IVUS interrogation.
* Baseline IVUS interrogation determined to be unacceptable by the Atherosclerosis Imaging Core Laboratory.
* ST-segment elevation myocardial infarction (STEMI) within the last 90 days
* Clinically significant heart disease which, in the opinion of the Investigator, is likely to require CABG, PCI cardiac transplantation, surgical or percutaneous valve repair, and/or replacement following index IVUS imaging (does not apply to PCI that occurs as a result of initial screening angiogram and completed prior to index IVUS imaging).
* New York Heart Failure Association Class III or IV heart failure or last known left ventricular ejection fraction <30%.
* Coronary artery bypass surgery <6 weeks prior to the qualifying IVUS.
* Cardiac arrhythmia within 3 months prior to randomization that is not controlled by medication.
* Uncontrolled severe hypertension: systolic blood pressure >180 millimeters of mercury (mmHg) or diastolic blood pressure >110 mmHg prior to randomization despite anti-hypertensive therapy.
* Poorly controlled diabetes mellitus and a hemoglobin A1c (HbA1c) >10.0% prior to randomization.
* Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or alanine aminotransferase, aspartate aminotransferase elevation >2 x ULN or total bilirubin elevation >1.5 x ULN at screening confirmed by a repeat measurement at least one week apart.
* Fasting triglyceride value >400 milligrams/deciliter (mg/dL).
* Impaired kidney function defined as calculated glomerular filtration rate <60 mL/minute by estimated glomerular filtration rate. In addition, participants with a 0.3 mg/dL or 25% increase in serum creatinine in the initial 3 to 5 days following angiography will be excluded from the study.
* Serious comorbid disease in which the life expectancy of the participant is shorter than the duration of the trial (such as, acute systemic infection, cancer, or other serious illnesses). This includes all cancers with the exception of treated basal-cell carcinoma occurring >3 years before screening.
* Body weight >120 kg.
* Females who are pregnant or nursing, or who are of childbearing potential and unwilling to use at least 2 methods of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal litigation). Women who are >2 years postmenopausal defined as ≥1 year since last menstrual period and are <55 years old with a negative pregnancy test within 24 hours of randomization or surgically sterile are exempt from this exclusion.
* Males who are unwilling to use an acceptable method of birth control during the entire study period (such as, condom with spermicide).
* Previous participation (enrollment and randomization) in this study or any preceding study with ETC-216 (predecessor compound of MDCO-216), MDCO-216, or similar investigational medicines containing apolipoprotein A-I (ApoA-I) proteins.
* Known allergy to the phospholipid or any other component of the investigational product (dimeric recombinant ApoA-IM, 1-palmitoyl-2-oleoyl-sn-glycero-3-phosphocholine, or mannitol and sucrose in phosphate buffer).
* Treatment with other investigational medicinal products or devices within 30 days or 5 half˗lives, whichever is longer.
* Known history of alcohol and/or drug abuse.
* Use of other investigational medicinal products or devices during the course of the study, excluding Post-Marketing Registries.
* Any condition that according to the investigator could interfere with the conduct of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2016-10-26 (Actual); Study Completion 2016-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nicholls, MBSS, PhD, Principal Investigator — South Australian Health & Medical Research Institute (SAHMRI) in Adelaide, Australia
Locations (20):
- Canada (3):
  - London
  - Québec
  - Winnipeg
- Czechia (3):
  - Brno
  - Hradec Králové
  - Prague
- Hungary (2):
  - Budapest
  - Szeged
- Netherlands (4):
  - Alkmaar
  - Amsterdam
  - Nijmegen
  - Venlo
- Poland (8):
  - Bielsko-Biala
  - Chrzanów
  - Dąbrowa Górnicza
  - Katowice
  - Kędzierzyn-Koźle
  - Krakow
  - Tychy
  - Warsaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nicholls SJ, Puri R, Ballantyne CM, Jukema JW, Kastelein JJP, Koenig W, Wright RS, Kallend D, Wijngaard P, Borgman M, Wolski K, Nissen SE. Effect of Infusion of High-Density Lipoprotein Mimetic Containing Recombinant Apolipoprotein A-I Milano on Coronary Disease in Patients With an Acute Coronary Syndrome in the MILANO-PILOT Trial: A Randomized Clinical Trial. JAMA Cardiol. 2018 Sep 1;3(9):806-814. doi: 10.1001/jamacardio.2018.2112. PMID 30046837

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who were screened, enrolled, randomized, received at least one infusion of study drug, and who had an evaluable Baseline and Follow-up intravascular ultrasound (IVUS) assessment were included in the modified intent-to-treat (mITT) population (primary/secondary analyses).
Groups:
- MDCO-216: 20 milligrams/kilogram (mg/kg) of MDCO-216 administered intravenously (IV) as a 360 milliliter (mL) infusion over 2 hours on Days 1, 8, 15, 22, and 29
Period: Overall Study
Arm/Group | MDCO-216 | Placebo
Started | 59 | 67
Received at Least 1 Dose of Study Drug (Randomized participants included in the Safety population.) | 58 | 64
mITT Population | 52 | 61
Completed | 53 | 62
Not Completed | 6 | 5
Not completed — Protocol Deviation (Not Dosed) | 1 | 3
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Did Not Return for Study Visits | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one infusion of study drug.
Groups:
- MDCO-216: 20 mg/kg of MDCO-216 administered IV as a 360 mL infusion over 2 hours on Days 1, 8, 15, 22, and 29
- Placebo: 360 mL of placebo (0.9% NaCl solution) infusion, IV, over 2 hours on Days 1, 8, 15, 22, and 29
- Total: Total of all reporting groups
Arm/Group | MDCO-216 | Placebo | Total
Number analyzed (Participants) | 58 | 64 | 122
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (10.6) | 61.4 (10.3) | 61.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 45 | 48 | 93
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 56 | 63 | 119
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 3 | 6
  Czech Republic | 3 | 2 | 5
  Hungary | 6 | 8 | 14
  Netherlands | 8 | 8 | 16
  Poland | 38 | 43 | 81

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Percent Atheroma Volume (PAV) At Day 36
Description: Change from Baseline to Day 36 post-randomization in PAV in a targeted (imaged) coronary artery for all anatomically comparable slices, as determined by IVUS. The change is calculated by subtracting the value at Baseline from the value at Day 36, with positive numbers to represent increases and negative numbers to represent decreases. Change in PAV was analyzed using an analysis of covariance (ANCOVA) model that included Baseline PAV as a covariate and treatment group as factor. Least Squares (LS) mean was adjusted for stratification factors of country and prior statin use.
Time Frame: Baseline, Day 36
Population: mITT population included all participants who were screened, enrolled, randomized, received at least one infusion of study drug, and who had an evaluable Baseline and Follow-up IVUS assessment.
Measure: Least Squares Mean (Standard Error); unit: change in percent
Arm/Group | MDCO-216 | Placebo
Number analyzed (Participants) | 52 | 61
change in percent | -0.21 (0.386) | -0.94 (0.382)
Statistical Analysis 1: Comparison: MDCO-216 vs Placebo; Test type: Superiority; p = 0.0738, ANCOVA — Baseline parameter value as a covariate and treatment group as factor, adjusting for country and prior statin use; LS mean difference = 0.73, 95% CI 2-sided [-0.07 to 1.52]

2. Secondary Outcome: Change From Baseline In Total Atheroma Volume (TAV) At Day 36
Description: Change from Baseline to Day 36 post-randomization in normalized TAV in a targeted (imaged) coronary artery for all anatomically comparable slices, as determined by IVUS. The change is calculated by subtracting the value at Baseline from the value at Day 36, with positive numbers to represent increases and negative numbers to represent decreases. Change in TAV was analyzed using an analysis of covariance (ANCOVA) model that included Baseline TAV as a covariate and treatment group as factor. LS mean was adjusted for stratification factors of country and prior statin use.
Time Frame: Baseline, Day 36
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: cubic millimeter (mm^3)
Arm/Group | MDCO-216 | Placebo
Number analyzed (Participants) | 52 | 61
cubic millimeter (mm^3) | -6.33 (3.425) | -7.89 (3.354)

3. Secondary Outcome: Change From Baseline In TAV For The 10 Millimeters (mm) Subsegment With The Greatest Disease Burden At Day 36
Description: Change in TAV from Baseline to Day 36 post-randomization of the most diseased 10-mm subsegment, as determined by IVUS. The change is calculated by subtracting the value at Baseline from the value at Day 36, with positive numbers to represent increases and negative numbers to represent decreases. Change in TAV was analyzed using an analysis of covariance (ANCOVA) model that included Baseline TAV for the most diseased 10-mm subsegment as a covariate and treatment group as factor. LS mean was adjusted for stratification factors of country and prior statin use.
Time Frame: Baseline, Day 36
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm^3
Arm/Group | MDCO-216 | Placebo
Number analyzed (Participants) | 52 | 61
mm^3 | -2.16 (1.809) | -1.74 (1.908)

4. Secondary Outcome: Participants With Regression Of Coronary Atherosclerosis As Measured By A PAV Change Greater Than 2 Standard Deviations Of Test-Retest Measurement Variability
Description: The number of participants with regression of coronary atherosclerosis is presented. For this Outcome Measure, the regression of coronary atherosclerosis is defined as a reduction in PAV from Baseline to Day 36 of greater than 2 standard deviations of the test-retest variability.
Time Frame: Baseline through Day 36
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | MDCO-216 | Placebo
Number analyzed (Participants) | 52 | 61
participants | NA — Test-retest requires IVUS to be done twice at the same time point and retest IVUS was not done. | NA — Test-retest requires IVUS to be done twice at the same time point and retest IVUS was not done.

5. Secondary Outcome: Participants With Regression Of Coronary Atherosclerosis As Measured By A PAV Change <0
Description: The number of participants with regression of coronary atherosclerosis is presented. For this Outcome Measure, the regression of coronary atherosclerosis is defined as a change in PAV from Baseline to Day 36 of less than zero.
Time Frame: Baseline through Day 36
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | MDCO-216 | Placebo
Number analyzed (Participants) | 52 | 61
Participants | 29 | 41

ADVERSE EVENTS:
Time Frame: Up to 59 days (±2 days) post randomization
Arm/Group | MDCO-216 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/64
Serious Adverse Events (participants affected / at risk) | 10/58 | 7/64
Other Adverse Events (participants affected / at risk) | 24/58 | 12/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MDCO-216 (N=58) | Placebo (N=64)
Angina unstable (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 3 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Vessel puncture site haemorrhage (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Echocardiogram abnormal (Investigations) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MDCO-216 (N=58) | Placebo (N=64)
Anaemia (Blood and lymphatic system disorders) | 3 | 4
Bradycardia (Cardiac disorders) | 3 | 1
Vessel puncture site haematoma (General disorders) | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 2
Gout (Metabolism and nutrition disorders) | 2 | 0
Dizziness (Nervous system disorders) | 4 | 1
Headache (Nervous system disorders) | 4 | 1
Insomnia (Psychiatric disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 4 | 2
Hypertension (Vascular disorders) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No